CLINICAL TRIAL: NCT02041676
Title: Evaluating the Impact of Chest Physiotherapy Technique Increasing Inspiratory Flow on Weaning From Non Invasive Ventilation (KVNI) Pilot Study
Brief Title: Chest Physiotherapy Technique Increasing Inspiratory Flow on Weaning From Non Invasive Ventilation
Acronym: KVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K 110701; A0007936 (Other: AP-HP)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-04

CONDITIONS: Neonatal Respiratory Distress Syndrome; Intubation, Intratracheal
Keywords: Chest; Physiotherapy; Increased Inspiratory Flow Technique; Prematurity; Non Invasive Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: chest physiotherapy technique (Experimental): Chest physiotherapy technique increasing inspiratory flow (IIF) 3 times per day
  Interventions: Procedure: Chest physiotherapy
- 2: Usual surveillance (Active Comparator): Usual surveillance of the non invasive ventilation
  Interventions: Procedure: Usual surveillance

INTERVENTIONS:
Procedure: Chest physiotherapy
  Other Names: Increased inspiratory flow technique (IIF)
  Arms: 1: chest physiotherapy technique
Procedure: Usual surveillance — Usual surveillance of the non invasive ventilation without chest physiotherapy.
  Arms: 2: Usual surveillance

SUMMARY:
The main objective is to show by a randomised controled therapeutic trial comparing in two parallel open arms ( 50 infants x 2 = 100 infants) that the technique IIF decreases the duration of non invasive respiratory support in the group treated by chest physiotherapy as compared to the control group. The secondary objectives are to evaluate the duration of oxygen dependence, the duration of hospitalisation and the proportional advent of bronchopulmonary dysplasia.

These study will be conducted in patients less than 32 weeks post menstrual age, eutrophic, treated by non invasive respiratory support after weaning off from mechanical endotracheal ventilation benefitting form a social security system and for whom the appropriate parental authority are non opposed.

DETAILED DESCRIPTION:
The treatment evaluated is the contribution of the chest physiotherapy technique of increasing the inspiratory flow (IIF) administered 3 times per day for a duration of 3 to 10 minutes according to the tolerance of the infant and interrupted if required by periods of rest. This technique utilises the exclusive nasal respiration and the increased thoracic compliance of the premature infant. The physiotherapy practiced engenders a progressive increase in the inspiratory flow until the physiological limits of the infant (expired volume and clinical tolerance). After having assured that the system is well in place, during the following inspiration we close the infant's mouth in a manner to add the following two simultaneous parameters of ventilation: forced inspiration and the PEP delivered by the ventilator. Regarding the Bi-phasic Positive Airway Pressure system of non invasive ventilation which is triggered by a movement captor placed on the skin of the lower thoracic cage, the physiotherapist will generate a first forced inspiration by following the respiratory rhythm of the infant. The infant will thus trigger the inspiratory aid of his machine simultaneously with the PEP delivered and the forced provoked inspiration.The respiratory rate of the infant can however be underestimated by the machine as it may not detect the ineffective respiratory efforts. The physiotherapy session shall be carried out by a physiotherapist of the service trained in this technique assisted by a nurse and the treatment shall start in the 24 hours following extubation/ weaning off form mechanical ventilation. The evaluation of clinical improvement will be done on a daily basis and the mode of non invasive respiratory support adapted accordingly. The objective of the project is to show that chest physiotherapy permits to decrease the duration of non invasive ventilation in the treatment group as compared to a control group without the above treatment ( this group will receive the usual care without the chest physiotherapy after extubation). Along with the expected diminution of the duration of non invasive respiratory support , we will also evaluate the efficiency of the IIF technique on the duration of oxygen dependence, the duration of hospitalisation of the premature infant on the special care unit, the proportion of infants diagnosed as having bronchopulmonary dysplasia at 36 weeks post menstrual age as established by the WALSH test as well as the presence of atelectasis on the chest X ray done within the 7 days following extubation. Eventual nociceptive effect will be evaluated by a pain score realised during the session.

This is a randomised controled therapeutic trial comparing two open parallel groups:

* A treatment group benefitting from the chest physiotherapy technique increasing inspiratory flow (IIF) 3 times per day along with the usual surveillance carried out under non invasive ventilation.
* A control group having the usual surveillance carried out under non invasive ventilation without any chest physiotherapy.

The research shall be carried out in one center. A draw to assign or not to the treatment group will be carried out by the physiotherapist present after having received the eligibility for the infant. The randomisation will be done by the physiotherapist with the aid of the electronic database CLEANWEB according to a list of pre established balanced randomisation ( size of the blocks not divulged to the investigators or the physiotherapists) after verification of the criteria of inclusion and information and explanation of the protocol to the parents.

Duration of inclusion: 24 months Duration of participation of each infant: 4 months maximum of treatment with follow up till discharge.

Duration of the research: 28 months Randomisation shall be done in the 24 hours following extubation. At all times the investigator can interrupt the study prematurely for a medical or administrative reason. In all cases the early termination will be done only after mutual discussion and appropriate documentation of the motives ( for example a letter of abandon for the investigator) and the investigator will inform the CPP.

If they want, the parental authority holders can at all times opt against the participation of their child in the study. In that case unless specifically desired otherwise, the data obtained during the inclusion of their child will be analysed This withdrawal from the study will not change the quality of the clinical management of their infant.

A termination of the study can be considered in case of insufficient recruitment, unresolved technical problems, expressed desire of the investigator or repeated and unjustified violation of the protocol.

In the setting of pathologies which might put at stake the vital prognostic of the patients a Surveillance Committee has been established to be able to:

* Follow the distribution of these events in the two arms of the study to make sure that there is no imbalance between the two.
* Make appropriate recommendations if need be (Eg: modification of the protocol ; continuation, suspension or early termination of the study etc. )"

ELIGIBILITY:
Inclusion Criteria:

* Infants < 32 weeks post menstrual age (corrected gestational age) and eutrophic on the AUDIPOG charts
* Patients with non invasive ventilation/ respiratory support following weaning from mechanical endo tracheal ventilation.
* Information letter given to the appropriate parental authority.
* Prior medical evaluation.
* Affiliation with a social security system.

Exclusion Criteria:

* Pneumothorax, emphysema, reintubation within 24 hours.
* Small for gestational age as defined by a birth weight < 10th percentile on the AUDIPOG charts.
* Intraventricular hemorrhage grade 3 and 4 (VOLPE's classification- (32-33))
* Thrombopenia (Platelet count < 80 000/mm3)
* Malformative syndromes

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of days of non invasive respiratory support post extubation | Data noted till discharge from special care (baby ) unit (4 months)

SECONDARY OUTCOMES:
Duration of oxygen dependence. | Data noted till discharge from special care (baby ) unit (4 months)
Duration of hospitalisation of the premature infant on the special care unit | 4 months
bronchopulmonary dysplasia as established by the WALSH test as well as the presence of atelectasis on the chest X ray done within the 7 days following extubation | at 36 weeks post menstrual age
Pain score realised during the session | until 4 months
  Eventual nociceptive effect

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Demont, Study Chair — Assistance Publique - Hôpitaux de Paris; Camille Roussel, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Antoine Béclère Hospital, Clamart, France

IPD SHARING:
Plan to Share IPD: No